CLINICAL TRIAL: NCT02144389
Title: Effects of Arachidonic Acid Supplementation on Schistosomiasis Mansoni Infection in Egyptian School Children
Brief Title: Arachidonic Acid Treatment Against Schistosomiasis Infection in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DSM Nutritional Products, Inc. (Industry)
Collaborators: National Liver Institute, Egypt (Other); Cairo University (Other); High Institute of Public Health, Egypt (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2012-1054
Record Dates: First submitted 2014-05-16; First posted 2014-05-22 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2014-05

CONDITIONS: Schistosomiasis; Bilharzia
Keywords: Arachidonic acid; Bilharzia; Mansoni; Schistosomiasis; Polyunsaturated fatty acid
MeSH Terms: conditions — Schistosomiasis | interventions — Praziquantel; Drugs, Generic; Arachidonic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Praziquantel (PZQ) (Active Comparator): A single dose of praziquantel (40 mg/kg) was administered orally on day-1 only, and after 7 days, 1 g of corn oil/soybean oil (50%/50%), for 15 consecutive days of school.
  Interventions: Drug: Praziquantel (PZQ)
- Arachidonic acid (ARA) (Experimental): A single daily dose of 1 g microbial arachidonic acid-rich oil administered orally for 15 consecutive days of school.
  Interventions: Dietary Supplement: Arachidonic acid (ARA)
- PZQ + ARA (Experimental): A single dose of PZQ (40 mg/kg) was administered orally on day-1 only, and after 7 days, followed the next day by 1 g of microbial ARA-rich oil, administered orally as a single dose on 15 consecutive days of school.
  Interventions: Dietary Supplement: PZQ+ARA

INTERVENTIONS:
Drug: Praziquantel (PZQ) — 40 mg/kg, a single dose, administered orally
  1 g of corn/soybean oil (50%/50%), administered orally
  Other Names: Praziquantel (generic); Biltricide; trematodicide
  Arms: Praziquantel (PZQ)
Dietary Supplement: Arachidonic acid (ARA) — ARA (40% of total fatty acid)
  Other Names: ARASCO; Microbial arachidonic acid-rich oil
  Arms: Arachidonic acid (ARA)
Dietary Supplement: PZQ+ARA — A single dose of PZQ administered seven days in advance of initial treatment with ARA.
  Other Names: ARASCO; praziquantel
  Arms: PZQ + ARA

SUMMARY:
Randomized Controlled Trial:

The investigational materials used in this trial were administered to subjects each day by trained clinicians.

Primary Objectives:

* assess the effect of dietary supplementation with arachidonic acid on the cure rates for Schistosomiasis mansoni with and without concomitant treatment with praziquantel.
* assess the safety of dietary supplementation using arachidonic acid in children with clinically confirmed schistosomiasis mansoni infection.

Secondary objective:

* to measure changes in total phospholipids in plasma.

ELIGIBILITY:
Inclusion Criteria:

* consent from parent or legal guardian
* clinically confirmed schistosomiasis

Exclusion Criteria:

* not infected with schistosomiasis
* less than 6 or greater than 15 years of age

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 335 (Actual)
Dates: Start 2013-01; Primary Completion 2013-07 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Percent egg reduction | 4 weeks after end of 1 day PZQ treatment
  Stool samples were collected from each child on three consecutive days to determine egg counts per gram of stool.

SECONDARY OUTCOMES:
Biochemical and hematological parameters | Three days after a 15-day ARA supplementation
  Blood samples were collected using 4 vacutainer tubes. Serum was used to measure enzyme markers of liver and kidney functions. Coagulation tests included prothrombin- and activated thromboplastin times were measured using citrated blood. Complete hematological profiles were obtained using EDTA-anticoagulated blood samples.
Total plasma phospholipids | Three days after 15-day ARA supplementation.
  Blood samples (10 ml) were collected 2-3 days before the start of treatment, and 3 days after completion of treatment with ARA or PZQ+ARA for analysis of the phospholipids in plasma.

CONTACTS AND LOCATIONS:
Overall Officials: Rashika El Ridi, Principal Investigator — Cairo University; Sahar Selim, Ph.D., Study Director — National Liver Institute, Menoufiya University; Rashida Barakat, Ph.D., Study Director — High Institute of Public Health, Alexandria University
Locations (3):
- Egypt (3):
  - National Liver Institute, Menoufiya University,, Shebin El-Kom, Monufia Governorate
  - Tropical Health Department, High Institute of Public Health, Alexandria University, Alexandria
  - Cairo University, Cairo

REFERENCES:
- [Derived] Barakat R, Abou El-Ela NE, Sharaf S, El Sagheer O, Selim S, Tallima H, Bruins MJ, Hadley KB, El Ridi R. Efficacy and safety of arachidonic acid for treatment of school-age children in Schistosoma mansoni high-endemicity regions. Am J Trop Med Hyg. 2015 Apr;92(4):797-804. doi: 10.4269/ajtmh.14-0675. Epub 2015 Jan 26. PMID 25624403